CLINICAL TRIAL: NCT01205633
Title: Multi-center Registry for CCSVI Testing and Treatment
Acronym: CCSVI
Status: Suspended | Type: Observational
Why Stopped: 9/12/12 FDA stopped enrollment pending device exemption(IDE)application.
Sponsor: Hubbard Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CCSVI Registry
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: CCSVI; Chronic Cerebrospinal Venous Insufficiency; Venous Malformations of CNS Draining Veins
Keywords: neurodegenerative disease; neurovascular disease; fatigue; Hubbard Foundation; angioplasty
MeSH Terms: conditions — Neurodegenerative Diseases; Fatigue

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CNS draining vein abnormalities
  Interventions: Procedure: venous angioplasty

INTERVENTIONS:
Procedure: venous angioplasty — catheter venous angioplasty via femoral vein approach

SUMMARY:
Patients suspected of CCSVI (chronic cerebrospinal venous insufficiency) may be tested and if appropriate treated with catheter venoplasty by an interventional radiologist in their local community who has been credentialled either by the local hospital's IRB or a national IRB if the procedure is done in an outpatient facility. Catheter angioplasty is a long-established and accepted medical procedure, patients' insurance should but may not cover the testing or treatment.

DETAILED DESCRIPTION:
more to follow

ELIGIBILITY:
Inclusion Criteria:

Referral by patients primary treating physician for suspected CCSVI

Exclusion Criteria:

Abnormal kidney function Allergy to either or both of the imaging contrast agents Pacemaker or other implantable device Ferrous metal in or on the body Claustrophobia Pregnancy

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of obstructions in the veins draining the central nervous system which may adversely affect CNS function
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Short-Form 36 (SF36) Quality of Life Instrument | Baseline and at 1, 6 and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: David R Hubbard, M.D., Study Chair — Hubbard Foundation
Locations (9):
- United States (9):
  - Vascular Access Center of Downey, Downey, California
  - North County Radiology, Oceanside, California
  - Vascular Access Care of Atlanta, Atlanta, Georgia
  - Columbia endovascular Associates, New York, New York
  - Valley Endovascular Associates, Poughkeepsie, New York
  - Dayton Interventional Radiology, Dayton, Ohio
  - Utah Valley Interventional Associates, Provo, Utah
  - Utah Vascular Clinic, Salt Lake City, Utah
  - Vascular Access Center of Seattle, Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.hubbardfoundation.org